CLINICAL TRIAL: NCT01642082
Title: A Phase II Evaluation of Dalantercept, a Novel Soluble Recombinant Activin Receptor-Like Kinase 1 (ALK-1) Inhibitor Receptor-Fusion Protein, in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Dalantercept in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0229N; NCI-2012-01986 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0229N; CDR0000736764; GOG-0229N (Other: NRG Oncology); GOG-0229N (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2012-07-15; First posted 2012-07-17 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2017-05

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Mixed Adenocarcinoma; Endometrial Mucinous Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Squamous Cell Carcinoma; Endometrial Transitional Cell Carcinoma; Endometrial Undifferentiated Carcinoma; Recurrent Uterine Corpus Carcinoma
MeSH Terms: interventions — ALK1-Fc fusion protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dalantercept) (Experimental): Patients receive dalantercept SC on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dalantercept; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Dalantercept — Given SC
  Other Names: ACE-041; Activin Receptor-like Kinase 1 Inhibitor ACE-041; ALK1-Fc Fusion Protein ACE-041
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well dalantercept works in treating patients with endometrial cancer that has come back or is persistent. Dalantercept may stop the growth of endometrial cancer by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients with persistent or recurrent endometrial cancer who survive progression-free for at least 6 months and the proportion of patients who have objective tumor response (complete or partial), treated with dalantercept (ACE-041).

II. To determine the nature and degree of toxicity of dalantercept in this cohort of patients.

SECONDARY OBJECTIVES:

I. To estimate progression-free survival (PFS) and overall survival (OS) of patients with persistent or recurrent endometrial cancer treated with dalantercept.

TERTIARY OBJECTIVES:

I. To measure the expression of vascular endothelial growth factor (VEGF), fibroblast growth factor (FGF), platelet-derived growth factor (PDGF), transforming growth factor-beta (TGF-β), activin receptor-like kinase 1 (ALK1), endoglin (CD105), and other markers via immunohistochemistry (IHC) and determine if there is correlation between expression and clinical response to treatment.

II. To determine the correlation between ALK1 gene expression, other markers, and clinical response to treatment.

III. To determine the correlation between concentration of VEGF, bone morphogenetic protein 9 (BMP9), bone morphogenetic protein 10 (BMP10), and ALK1 in pre-cycle 1 plasma using an enzyme-linked immunosorbent assay (ELISA), and clinical response to treatment.

IV. To correlate somatic mutations in candidate genes with response to therapy.

OUTLINE:

Patients receive dalantercept subcutaneously (SC) on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent endometrial carcinoma; histologic confirmation of the original primary tumor is required

  * Patients with the following histologic epithelial cell types are eligible: Endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, and transitional cell carcinoma
* All patients must have measurable disease; measurable disease is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1) as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be > 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST version 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III protocol or rare tumor protocol for the same patient population
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2; patients who have received two prior regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
  * Any other prior therapy directed at the malignant tumor, including chemotherapy and immunologic agents, must be discontinued at least three weeks prior to registration; any investigational drug must be discontinued at least 30 days prior to registration
  * Any prior radiation therapy must be discontinued at least four weeks prior to registration
  * At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: laparotomy, laparoscopy); there is no delay in treatment for minor procedures (e.g., central venous access catheter placement)
* Prior therapy

  * Patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma. Initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen
  * Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease
  * Patients must have NOT received any non-cytotoxic (biologic or targeted) agent(s) for management of recurrent or persistent disease; prior non-cytotoxic (biologic or targeted) agent(s) is allowed as part of initial treatment; prior hormonal therapy is allowed, but must be discontinued at least one week prior to registration
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcL
* Platelets greater than or equal to 100,000/mcL
* Hemoglobin greater than or equal to 9 g/dL
* Creatinine less than or equal to 1.5 times institutional upper limit normal (ULN)
* Sodium greater than or equal to 130 mEq/L (Common Terminology Criteria for Adverse Events [CTCAE] v. 4, grade 0 or 1)
* Urine protein should be screened by urinalysis; if protein is 2+ or higher, 24-hour urine protein should be obtained and the level should be < 1,000 mg (< 1.0 g/24 hrs) for patient enrollment
* Bilirubin less than or equal to 1.5 times ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 3 times ULN
* Alkaline phosphatase less than or equal to 3 times ULN
* Albumin greater than or equal to 3 (CTCAE v. 4, grade 0 or 1)
* Prothrombin time (PT) such that international normalized ratio (INR) is less than or equal to 1.5 times ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin)
* Partial thromboplastin time (PTT) less than or equal to 1.5 times ULN
* Left ventricular ejection fraction (LVEF) greater than 50% (measured by echocardiogram or MUGA [multi-gated acquisition] scan)
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception

Exclusion Criteria:

* Patients who have had prior therapy with dalantercept or other inhibitor of the ALK1 pathway
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with history or evidence upon physical exam of central nervous system disease (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, or any brain metastases or leptomeningeal disease
* Serious or non-healing wound, ulcer, or bone fracture
* History of abdominal fistula or anastomotic leak, gastrointestinal perforation, or intra-abdominal abscess within 6 months of registration
* Patients requiring parenteral hydration or parenteral/total parenteral nutrition
* No patients with:

  * Active bleeding (e.g., active hemoptysis, defined as bright red blood of greater than or equal to ½ teaspoon [2.5 ml] in any 24-hour period) within 2 weeks prior to registration or gastrointestinal bleeding within 3 months prior to registration
  * Hereditary hemorrhagic telangiectasia (HHT)
  * Platelet function abnormality
  * Autoimmune or hereditary hemolysis
  * Coagulopathy, or
  * Tumor involving major vessels (defined as any lesion invading or abutting the wall [i.e., no fat plane evident] of major blood vessels as assessed by CT or MRI)
* Patients receiving treatment with full-dose aspirin (325 mg oral daily), clopidogrel (Plavix), or dabigatran (Pradaxa)
* Patients with peripheral edema greater than or equal to grade 1 within 4 weeks of registration
* No patients with clinically significant cardiovascular disease:

  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg despite antihypertensive medications
  * Evidence of hypertrophic cardiomyopathy
  * New York Heart Association (NYHA) class II or greater congestive heart failure (CHF)
  * Any of the following within 6 months prior to study registration:

    * Bypass surgery
    * Stent placement
    * Myocardial infarction
    * Acute coronary syndrome/unstable angina
    * Hospitalization for congestive heart failure (CHF)
  * Serious cardiac arrhythmia requiring medication; this does not include asymptomatic atrial fibrillation with controlled ventricular rate
  * Prolonged QTc interval > 450 ms
  * Prior anthracycline cumulative dose > 450 mg/m^2
* Patients who are pregnant or nursing
* History of syndrome of inappropriate antidiuretic hormone secretion (SIADH)
* Patients who have undergone a therapeutic paracentesis within 4 weeks of registration
* Known history of positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg), or HBV core antibody, or human immunodeficiency virus (HIV) antibody results
* History of severe (National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] v.4.0 >= grade 3) allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or excipients (10 mM Tris buffered saline) in the investigational agent
* Clinically significant active pulmonary risk including pulmonary hypertension, pulmonary embolism, or history of pulmonary edema

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Makker, Principal Investigator — NRG Oncology
Locations (30):
- United States (30):
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Florida Hospital Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Union Hospital of Cecil County, Elkton, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford NCI Community Oncology Research Program of the North Central Plains, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Pacific Gynecology Specialists, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients underwent disease evaluation with baseline CT of the chest, abdomen and pelvis. After obtaining informed consent and verification of eligibility, patients were enrolled and treatment initiated.
Groups:
- Dalantercept: Dalantercept 1.2 mg/kg (maximum starting dose of 120 mg) subcutaneously once every three weeks. One cycle is defined as three weeks.
  Patients weighing more than 100 kg start treatment at 120 mg, and if dalantercept is tolerated for 2 cycles (i.e. toxicities are tolerable, less than grade 2 and resolved), the patient can be dose escalated to dosing based on actual body weight.
  A CT of the chest, abdomen and pelvis to assess response by RECIST 1.1 is required every two cycles. Treatment was to continue until disease progression or adverse effects prohibit further therapy.
Period: Overall Study
Arm/Group | Dalantercept
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Dalantercept)
Number analyzed (Participants) | 28
Age, Customized [Number; unit: participants]
  40-49 | 1
  50-59 | 9
  60-69 | 13
  70-79 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Response was defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) and based on imaging done every other cycle. Responses can be either partial or complete. Per RECIST v1.1 target and non-target lesions are assessed by MRI or CT scan: Complete Response (CR), Disappearance of all target and non-target lesions and all lymph nodes must be < 10 mm in short axis; Partial Response (PR), >=30% decrease in the sum of the longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD.
Time Frame: Scans to assess response were done every other cycle for the first 6 months; every three months thereafter; and any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease. Responses must be confirmed.
Population: All eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dalantercept
Number analyzed (Participants) | 28
percentage of participants | 0 [0 to 10.1]

2. Primary Outcome: Treatment and Progression-free Survival at 6 Months
Description: Treatment and Progression-free Survival is defined as the duration alive from study entry until progression is documented, death or non-protocol treatment is initiated; whichever comes sooner. Progressive disease is defined as at least a 5 mm absolute increase and a 20% relative increase in the sum of measurable target lesions' longest dimensions relative to the smallest sum at baseline or on study or the appearance of new lesions or unequivocal progression of existing non-target lesions.
  Non-protocol treatment initiation prior to disease progression and prior to 6 months from study entry was counted as an event for treatment and progression-free survival at 6 months. Disease progression within 6 months of study entry or death within 6 months of study entry and prior to disease progression counts as an event for treatment and progression-free survival at 6 months.
Time Frame: CT scan or MRI were to assess progression every other cycle for the first 6 months; every three months thereafter; and any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease
Population: All eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dalantercept
Number analyzed (Participants) | 28
percentage of participants | 10.7 [3 to 25.4]

3. Secondary Outcome: Progression-free Survival at 6 Months
Description: Progression-free survival is defined as the duration alive from study entry until progression is documented or death, whichever comes sooner. Progressive disease is defined as at least a 5 mm absolute increase and a 20% relative increase in the sum of measurable target lesions' longest dimensions relative to the smallest sum at baseline or on study or the appearance of new lesions or unequivocal progression of existing non-target lesions.
  Disease progression within 6 months of study entry or death within 6 months of study entry and prior to disease progression counts as an event for progression-free survival at 6 months.
Time Frame: : CT scan or MRI were to assess progression every other cycle for the first 6 months; every three months thereafter; and any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease.
Population: All eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dalantercept
Number analyzed (Participants) | 28
percentage of participants | 17.9 [7.3 to 33.9]

4. Secondary Outcome: Duration of Progression-free Survival
Description: Progression-free survival is defined as the duration alive from study entry until progression is documented or death, whichever comes sooner. Progressive disease is defined as at least a 5 mm absolute increase and a 20% relative increase in the sum of measurable target lesions' longest dimensions relative to the smallest sum at baseline or on study or the appearance of new lesions or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 2
Population: All eligible and treated patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Dalantercept)
Number analyzed (Participants) | 28
months | 2.1 [1.4 to 3.2]

5. Secondary Outcome: Duration of Survival
Description: Duration of survival is defined as the duration alive from study entry until death or last contact.
Time Frame: Patients are followed every three months for the first two years and then every six months for the next three years.
Population: All eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Dalantercept
Number analyzed (Participants) | 28
months | 14.5 [7.0 to 17.5]

6. Secondary Outcome: Adverse Events (Primary Serious and All Other AEs)
Description: The frequencies of the maximum grade of any acute adverse event, regardless of attribution are reported during treatment and up to 30 days after stopping the study treatment are reported.
Time Frame: Every cycle of study treatment and after treatment for a maximum of 5 years from study entry
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v4.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 4.0
- Grade 2 (CTCAE v4.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 4.0
- Grade 3 (CTCAE v 4.0): Number of patients who experienced a grade 3 event using Common Terminology version 4.0
- Grade 4 (CTCAE v 4.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 4.0
- Grade 5 (CTCAE v 4.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 4.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v4.0) | Grade 2 (CTCAE v4.0) | Grade 3 (CTCAE v 4.0) | Grade 4 (CTCAE v 4.0) | Grade 5 (CTCAE v 4.0)
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28 | 28
Participants
  Anemia | 13 | 5 | 8 | 1 | 1 | 0
  Abdominal Distention | 24 | 2 | 2 | 0 | 0 | 0
  Abdominal Pain | 20 | 6 | 2 | 0 | 0 | 0
  Ascites | 24 | 0 | 2 | 2 | 0 | 0
  Constipation | 11 | 12 | 5 | 0 | 0 | 0
  Diarrhea | 22 | 5 | 1 | 0 | 0 | 0
  Gastric Hemorrhage | 27 | 0 | 0 | 0 | 0 | 1
  Nausea | 16 | 11 | 1 | 0 | 0 | 0
  Rectal Fistula | 27 | 0 | 0 | 1 | 0 | 0
  Rectal Hemorrhage | 26 | 2 | 0 | 0 | 0 | 0
  Vomiting | 19 | 8 | 0 | 1 | 0 | 0
  Edema Face | 26 | 1 | 1 | 0 | 0 | 0
  Edema Limbs | 11 | 15 | 2 | 0 | 0 | 0
  Fatigue | 4 | 17 | 6 | 1 | 0 | 0
  Prolonged activated partial thromboplastin time | 27 | 0 | 0 | 1 | 0 | 0
  Alkaline Phosphatase Increased | 22 | 4 | 2 | 0 | 0 | 0
  Creatinine Increased | 19 | 5 | 4 | 0 | 0 | 0
  Lymphocyte Count Decreased | 25 | 1 | 1 | 1 | 0 | 0
  Weight Loss | 24 | 2 | 2 | 0 | 0 | 0
  Anorexia | 24 | 2 | 2 | 0 | 0 | 0
  Dehydration | 26 | 0 | 2 | 0 | 0 | 0
  Hyperglycemia | 22 | 5 | 1 | 0 | 0 | 0
  Hypoalbuminemia | 19 | 4 | 4 | 1 | 0 | 0
  Hypoglycemia | 27 | 0 | 1 | 0 | 0 | 0
  Hypokalemia | 24 | 1 | 2 | 1 | 0 | 0
  Arthralgia | 24 | 4 | 0 | 0 | 0 | 0
  Back Pain | 19 | 4 | 4 | 1 | 0 | 0
  Myalgia | 25 | 3 | 0 | 0 | 0 | 0
  Dizziness | 26 | 2 | 0 | 0 | 0 | 0
  Headache | 15 | 13 | 0 | 0 | 0 | 0
  Neuralgia | 27 | 0 | 1 | 0 | 0 | 0
  Urinary Tract Obstruction | 27 | 0 | 0 | 1 | 0 | 0
  Dyspnea | 18 | 8 | 1 | 1 | 0 | 0
  Epistaxis | 24 | 4 | 0 | 0 | 0 | 0
  Pleural Effusion | 24 | 1 | 2 | 1 | 0 | 0
  Hypertension | 25 | 1 | 1 | 1 | 0 | 0
  Thromboembolic Event | 26 | 0 | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Every cycle of study treatment and after treatment for a maximum of 5 years from study entry
Description: The frequencies of the maximum grade of any serious adverse event or all other adverse events by category or specific term occurring during treatment and up to 30 days after stopping the study treatment are reported
Arm/Group | Dalantercept
Serious Adverse Events (participants affected / at risk) | 11/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalantercept (N=28)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Rectal Fistula (Gastrointestinal disorders) | 1 (1)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thromboembolic Event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalantercept (N=28)
Anemia (Blood and lymphatic system disorders) | 15
Ventricular Arrhythmia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hearing Impaired (Ear and labyrinth disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 2
Flashing Lights (Eye disorders) | 1
Eye Pain (Eye disorders) | 2
Blurred Vision (Eye disorders) | 3
Floaters (Eye disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 9
Abdominal Pain (Gastrointestinal disorders) | 8
Rectal Hemorrhage (Gastrointestinal disorders) | 2
Mucositis Oral (Gastrointestinal disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 12
Gastroparesis (Gastrointestinal disorders) | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 4
Pain (General disorders) | 3
Localized Edema (General disorders) | 1
Injection Site Reaction (General disorders) | 1
Edema Trunk (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 2
Edema Limbs (General disorders) | 17
Edema Face (General disorders) | 2
Fatigue (General disorders) | 24
Fever (General disorders) | 1
Wound Infection (Infections and infestations) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Soft Tissue Infection (Infections and infestations) | 1
Papulopustular Rash (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Weight Loss (Investigations) | 4
Weight Gain (Investigations) | 2
Lymphocyte Count Decreased (Investigations) | 3
Creatinine Increased (Investigations) | 9
Aspartate Aminotransferase Increased (Investigations) | 4
Alkaline Phosphatase Increased (Investigations) | 6
Alanine Aminotransferase Increased (Investigations) | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Peripheral Sensory Neuropathy (Nervous system disorders) | 5
Paresthesia (Nervous system disorders) | 4
Neuralgia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 13
Facial Nerve Disorder (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2
Urinary Tract Pain (Renal and urinary disorders) | 2
Urinary Frequency (Renal and urinary disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 2
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Urticaria (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Periorbital Edema (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2
Telangiectasia (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3
Thromboembolic Event (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No